CLINICAL TRIAL: NCT03420625
Title: Haemodynamic Effects of Different Mechanical Compression Devices and Neuromuscular Stimulation in the Lower Limb
Brief Title: Blood Flow Stimulation in the Lower Limbs by Application of Different External Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Principal Investigator, Karolinska University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SW2016-17-HEMOD
Record Dates: First submitted 2017-02-08; First posted 2018-02-05 (Actual); Results first posted 2019-02-12 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Venous Stasis; Deep Vein Thrombosis
Keywords: Intermittent Pneumatic Compression Devices; Electric Stimulation Therapy; Blood Flow Velocity; Hemodynamics
MeSH Terms: conditions — Varicose Ulcer; Venous Thrombosis

ARMS (4):
- Foot IPC (Active Comparator): Intermittent pneumatic compression in the foot using the A-V Impulse™, Covidien®, New Haven, CT, USA
  Interventions: Device: Foot IPC
- Rapid calf IPC (Active Comparator): Intermittent pneumatic compression in the calf using the VenaFlow® Elite, DJO Global, USA
  Interventions: Device: Rapid calf IPC
- Slow calf IPC (Active Comparator): Intermittent pneumatic compression in the calf using the Kendall SCD™ 700, Covidien, Medtronic, USA
  Interventions: Device: Slow calf IPC
- Calf NMES (Active Comparator): Neuromuscular electrical stimulation in the calf using the DJO,TM, CefarCompex Mi-Theta 500 stimulator
  Interventions: Device: Calf NMES

INTERVENTIONS:
Device: Foot IPC — Intermittent pneumatic compression in the foot using the A-V Impulse™, Covidien®, New Haven, CT, USA
  Other Names: Intermittent pneumatic compression in the foot
  Arms: Foot IPC
Device: Rapid calf IPC — Intermittent pneumatic compression in the calf using the VenaFlow® Elite, DJO Global, USA
  Other Names: Rapid Intermittent pneumatic compression in the calf
  Arms: Rapid calf IPC
Device: Slow calf IPC — Intermittent pneumatic compression in the calf using the Kendall SCD™ 700, Covidien, Medtronic, USA
  Other Names: Slow Intermittent pneumatic compression in the calf
  Arms: Slow calf IPC
Device: Calf NMES — Neuromuscular electrical stimulation in the calf using the DJOTM, CefarCompex Mi-Theta 500 stimulator
  Other Names: Calf neuromuscular electrical stimulation
  Arms: Calf NMES

SUMMARY:
In this study, four different devices which stimulate the blood in the lower extremities are used in ten healthy persons while measuring the blood flow with ultrasound. The aim is to study the haemodynamic effects in the lower extremities of each modality and also to compare those effects between the four modalities in order to identify those which most effective than the others.

DETAILED DESCRIPTION:
Three Intermittent Pneumatic Compression (IPC) devices were selected: Foot-IPC, rapid Calf-IPC and a slow, sequential Calf-IPC. A Neuromuscular Electrical Stimulation (NMES) device was also used in the calf. Blood flow measurements in the right popliteal vein of ten healthy individuals were performed using Doppler ultrasound before (control) and while using IPC or NMES. The blood flow parameters measured where: peak systolic velocity (cm/s), time-averaged mean velocity (cm/sec), volume flow (ml/min) and ejected volume per individual stimulus (ml). The tolerability of each device was also assessed using an analogue scale from zero to ten. Differences between modalities regarding the pattern as well as the absolute values of velocity and volume are being assessed. Power calculation: Recent studies showed that the peak venous velocity (PV) at baseline is around 11 cm/s and after applying foot-IPC the PV rises to 50 cm/s with a maximum standard deviation of 15 (Broderick et all, 2014). Thus, three patients per group would be required to detect a difference of 39 cm/s in PV (two-sided type-I error rate = 5%; power = 80%). To reach an even higher power we choose to include 10 patients in study, which resulted in a power of 99.7% for the above calculation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* pregnancy
* previous lower limb operation involving the vascular system
* current thromboprophylactic or thrombolytic therapy
* vascular abnormalities in the lower limbs
* cardiorespiratory or renal failure causing pitting oedema

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemodynamic Studies: Patients undergoing different interventions to promote venous return. Washout (1 hour) in between different interventions. Patients started in different orders with: "Foot IPC", "Rapid Calf IPC", "Slow Calf IPC" and "Calf NMES".
Period: Overall Study
Arm/Group | Hemodynamic Studies
Started | 10
Baseline (Venous flow in the popliteal vein during supine position) | 10
Foot IPC (Intermittent pneumatic compression of the foot using A-V Impulse™, Covidien®, New Haven, CT, USA) | 10
Rapid Calf IPC (Intermittent pneumatic compression of the calf using the VenaFlow® Elite, DJO Global, USA) | 10
Slow Calf IPC (Intermittent pneumatic compression of the calf using the Kendall SCD™ 700, Covidien, Medtronic, USA) | 10
Calf NMES (Neuromuscular electrical stimulation of the calf using the CefarCompex Mi-Theta 500 stimulator) | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hemodynamic Studies: Patients undergoing different stimulations of venous blood flow.
Arm/Group | Hemodynamic Studies
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 10

OUTCOME MEASURES:

1. Primary Outcome: Blood Flow - Peak Systolic Velocity (cm/Sec)
Description: With the use of Doppler Ultrasound Peak systolic velocity (cm/sec) is assessed in the popliteal vein.
Time Frame: up to one hour in total
Population: The interventions were performed sequentially on each participant as listed after baseline, in total 10 participants.
  One patient did not perform the Rapid calf IPC intervention
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Baseline: Venous blood flow during supine position
Arm/Group | Baseline | Foot IPC | Rapid Calf IPC | Slow Calf IPC | Calf NMES
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10
cm/s | 14.1 (3.42) | 29.5 (8.4) | 161.6 (47.8) | 39.0 (12.5) | 42.1 (14.9)

2. Primary Outcome: Blood Flow - Time-averaged Mean Velocity (cm/Sec)
Description: With the use of Doppler Ultrasound Time-averaged mean velocity (cm/sec) is assessed in the popliteal vein.
Time Frame: up to one hour in total
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Baseline: Blood flow during supine position
Arm/Group | Baseline | Foot IPC | Rapid Calf IPC | Slow Calf IPC | Calf NMES
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10
cm/s | 4.58 (1.18) | 6.53 (1.29) | 13.24 (6.35) | 7.12 (1.33) | 9.18 (2.30)

3. Primary Outcome: Blood Flow - Volume Flow (ml/Min)
Description: With the use of Doppler Ultrasound Volume flow (ml/min), is assessed in the popliteal vein.
Time Frame: up to one hour in total
Measure: Median (Standard Deviation); unit: ml/min
Arm/Group | Baseline | Foot IPC | Rapid Calf IPC | Slow Calf IPC | Calf NMES
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10
ml/min | 219 (104) | 309 (132) | 604 (303) | 345 (124) | 410 (184)

4. Primary Outcome: Blood Flow - Ejected Volume Per Individual Stimulus (ml)
Description: With the use of Doppler Ultrasound Ejected volume per individual stimulus (ml) is assessed in the popliteal vein.
Time Frame: up to one hour in total
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Baseline | Foot IPC | Rapid Calf IPC | Slow Calf IPC | Calf NMES
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10
ml | 5.5 (3.96) | 9.4 (4.0) | 19.8 (8.6) | 60.8 (22.2) | 13.6 (5.9)

5. Secondary Outcome: Tolerability to IPC and NMES According to Visual Analogue Scale 0-10
Description: All subjects will be asked to subjectively grade each modality according to how comfortable or uncomfortable it felt under the time was applied to the subject according to Visual Analogue Scale 0-10. The following description will be given to the subjects: 0 denotes the the modality was totally intolerable, 10 denotes that the modality is very pleasant to use and 5 denotes neither pleasant nor unpleasant feeling.
Time Frame: one minute
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Foot IPC | Rapid Calf IPC | Slow Calf IPC | Calf NMES
Number analyzed (Participants) | 10 | 9 | 10 | 10
units on a scale | 6.13 (1.36) | 6.3 (1.17) | 8.0 (1.07) | 3.3 (1.67)

ADVERSE EVENTS:
Time Frame: 8 hours during the baseline and intervention assessments.
Description: The interventions were performed sequentially on each participant after baseline, in total 10 participants.
  One patient did not perform the Rapid calf IPC intervention. Adverse events were registered during and after the application of these interventions.
  Specifically assessments of pain were made during the application of each intervention.
Arm/Group | Foot IPC | Rapid Calf IPC | Slow Calf IPC | Calf NMES
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foot IPC (N=10) | Rapid Calf IPC (N=9) | Slow Calf IPC (N=10) | Calf NMES (N=10)
Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) — Pain in the limb with cramping sensation when applying NMES. Comfortability scale (0-10). When patients scored 4 or less.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes